CLINICAL TRIAL: NCT05638828
Title: A Study of RD14-01 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shen Lin (Other)
Responsible Party: Sponsor-Investigator, Shen Lin, Professor, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD14-01-03
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor
Keywords: CAR-T Cell; ROR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cell injection (Experimental)
  Interventions: Drug: RD14-01 Cell injection

INTERVENTIONS:
Drug: RD14-01 Cell injection — RD14-01 Cell injection

SUMMARY:
This study will evaluate the safety and tolerability of RD14-01, a ROR1-targeted CAR T-cell therapy, in patients with ROR1+ advanced solid tumors.

DETAILED DESCRIPTION:
This single-arm, open-label, dose-escalation and dose-expansion study will evaluate the safety and tolerability of RD14-01, ROR1-targeting CAR T cells, in adults with ROR1+ advanced solid tumors. The dose-escalation phase will investigate 3 dose levels to the. The dose-expansion phase will enroll .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients with histologically or cytologically confirmed advanced solid tumor, who have progressive disease, have undergone systemic therapy for advanced disease, and for whom no standard therapy is available.
3. ROR1+ by central laboratory immunohistochemistry (IHC).
4. Adequate organ and marrow function.
5. At least one measurable lesion as per RECIST v1.1.
6. . Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Ability to understand and provide informed consent.

Exclusion Criteria:

1. Prior treatment with any agent targeting ROR1
2. Presence of active central nervous system (CNS) metastasis
3. Impaired cardiac function or clinically significant cardiac disease
4. Untreated or active infection at the time of screening or leukapheresis
5. HIV-positive, active acute or chronic HBV or HCV, or active tuberculosis
6. Untreated or active infection at the time of screening or leukapheresis
7. Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
DLT and MTD | up to 28 days
  Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD)
TEAEs | up to 12 months
  Adverse events (TEAEs) and incidence after the first infusion, treatment-related adverse events and incidence, adverse events of special concern (AESI) and incidence.

SECONDARY OUTCOMES:
ORR | up to 28 days
  Overall Response Rate (ORR) by RECIST, version 1.1
DOR | up to 12 months
  Duration of response (DOR)
PFS | up to 12 months
  Progression Free Survival(PFS)
OS | up to 12 months
  Overall Survival (OS)
Maximum concentration of RD14-01 (Cmax) in peripheral blood (PB) samples | up to 12 months
  Maximum concentration of RD14-01 (Cmax) in peripheral blood (PB) samples
Time to Cmax (Tmax) of RD14-01 in peripheral blood (PB) samples | up to 12 months
  Time to Cmax (Tmax) of RD14-01 in peripheral blood (PB) samples
Persistence of RD14-01 CAR T cells in peripheral blood samples | up to 12 months
  Persistence of RD14-01 CAR T cells in peripheral blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Prof. Dr., Principal Investigator — Peking University Cancer Hospital & Institute